CLINICAL TRIAL: NCT03989713
Title: Quizartinib and High-dose Ara-C Plus Mitoxantrone in Relapsed/Refractory AML With FLT3-ITD
Acronym: Q-HAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study turned out no longer feasible
Sponsor: Prof. Dr. Richard F Schlenk (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Richard F Schlenk, Head of NCT trials center and Clinical Trials Office Hematology/Oncology, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HeLeNe-18-03-#545
Record Dates: First submitted 2019-04-12; First posted 2019-06-18 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: AML According to WHO 2016 Classification (Except Acute Promyelocytic Leukemia) AND (Refractory to Induction Therapy OR Relapsed After First Line Treatment)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD-triggered arm (Experimental): 1. Salvage therapy: All patients are randomized upfront and receive one cycle Q-HAM salvage therapy. All patients achieving CR or CRi are allocated according to randomization to either MRD-triggered or prophylactic arm.
     (Duration: one cycle á 21 days followed by up to 3 weeks recovery period if needed, 22-42 days in total)
  2. Consolidation therapy: Patients receive one cycle of HAM and are further allocated based on the MRD-results assessed by flow cytometry with a cut of level of 0.1%: if the MRD is negative they remain in the MRD-triggered arm, whereas MRD positive patients cross over to the prophylactic arm.
     (Up to 2 cycles. Duration: two cycles á 28 days each followed by up to two weeks recovery period if needed, 56-84 days in total.)
  3. Observation: No treatment will be given in the MRD-triggered arm. (Duration: 48 weeks in total.)
  4. Safety follow-up and observational follow-up
  Interventions: Drug: MRD-triggered arm
- Prophylactic Arm (Experimental): 1. Salvage therapy: All patients are randomized upfront and receive one cycle Q-HAM salvage therapy. All patients achieving CR or CRi are allocated according to randomization to either MRD-triggered or prophylactic arm.
     (Duration: one cycle á 21 days followed by up to 3 weeks recovery period if needed, 22-42 days in total)
  2. Consolidation therapy: Patients may receive up to two cycle of Q-HAM. (Up to 2 cycles. Duration: two cycles á 28 days each followed by up to two weeks recovery period if needed, 56-84 days in total.)
  3. Maintenance therapy: Quizartinib will be given as single-agent therapy. The dose of quizartinib is aimed to be increased during maintenance therapy. (Up to 12 cycles. Duration: four times three cycles á 28 days, 48 weeks in total.)
  4. Safety follow-up and observational follow-up
  Interventions: Drug: Prophylactic Arm

INTERVENTIONS:
Drug: MRD-triggered arm — 1. Salvage therapy:
     Quizartinib: 40mg, p.o., Days: 4 - 21 Cytarabine: 18-60yrs: 3g/m² bid / >-60yrs: 1g/m² bid, i.v. 3h i.v. 3h, Days: 1,2,3; Mitoxantrone: 10mg, i.v. 30min: Days: 2,3;
  2. Consolidation therapy:
     Cytarabine: 18-60yrs: 3g/m² bid, i.v. 3h / >-60yrs: 1g/m² bid, i.v. 3h, Days: 1,2,3; Mitoxantrone: 10mg, i.v. 30min, Days: 2,3
  3. Observation therapy:
  No treatment
  Arms: MRD-triggered arm
Drug: Prophylactic Arm — 1. Salvage therapy:
     Quizartinib: 40mg, p.o., Days: 4 - 21 Cytarabine: 18-60yrs: 3g/m² bid / >-60yrs: 1g/m² bid, i.v. 3h i.v. 3h, Days: 1,2,3; Mitoxantrone: 10mg, i.v. 30min: Days: 2,3;
  2. Consolidation therapy:
     Quizartinib: 40mg, p.o., Days: 4 - 21 Cytarabine: 18-60yrs: 3g/m² bid, i.v. 3h / >-60yrs: 1g/m² bid, i.v. 3h, Days: 1,2,3; Mitoxantrone: 10mg, i.v. 30min, Days: 2,3;
  3. Maintenance therapy:
  Quizartinib: Cycle 1, Days 1-15: 40mg, p.o. and Day 16-28: 60mg, p.o.
  Arms: Prophylactic Arm

SUMMARY:
In this multicenter, upfront randomized phase II trial, all patients receive quizartinib in combination with HAM (high-dose cytarabine, mitoxantrone) during salvage therapy. Efficacy is assessed by comparison to historical controls based on the matched threshold crossing approach. During consolidation therapy (chemotherapy as well as allo-HCT) patients receive either prophylactic quizartinib therapy or MRD-triggered preemptive continuation therapy with quizartinib according to up-front randomization.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a clonal malignant disorder which is characterized by the expansion of leukemic blasts in the bone marrow and the peripheral blood, which goes along with a suppression of normal hematopoiesis including granulopoiesis, erythropoiesis and thrombocytopoiesis. The prognosis is largely determined by cytogenetic and molecular risk factors, age, performance status and antecedent myelodysplastic syndrome (MDS). With the exception of old and frail patients, most AML patients are eligible for intensive chemotherapy, which is given in curative intent consisting of induction and consolidation therapy. However, despite intensive therapy, the long-term outcome of AML patients remains poor, with less than 30% of patients achieving long lasting remission and even cure. This poor outcome is largely due to refractoriness to induction chemotherapy as well as relapses during and after completion of intensive induction and consolidation therapy. Regarding refractoriness, about 20-30% of AML patients under the age of 60 years and about 50% of older patients fail to attain complete remission (CR) following cytarabine plus anthracycline based standard induction therapy. In addition, patients having achieved CR are at a high risk of relapse, particularly within the first two years after completion of chemotherapy. Allogeneic hematopoietic cell transplantation (allo-HCT) is currently the only treatment strategy to offer the prospect of cure in relapsed/refractory (r/r)-AML; but outcome after allo-HCT is largely determined by the remission state before allo-HCT. With the aim to induce a CR before allo-HCT, salvage chemotherapy regimens are administered in r/r-AML. Typically, these salvage regimens are based on high dose cytarabine (HiDAC), which is frequently combined with either mitoxantrone (HAM regimen) or fludarabine plus idarubicin (idaFLA regimen). However, there is still no commonly accepted standard salvage regimen and overall CR rates remain low with less than one third of the patients achieving a CR. Apart from already known clinical unfavorable prognostic parameters in relapsed AML such as short first CR duration, older age and previous allo-HCT, FLT3-ITD has consistently been identified as an unfavorable molecular marker in both relapsed and refractory AML. Recently midostaurin has been approved by the FDA and EMA for the treatment of newly diagnosed AML with activating FLT3 mutations. But still roughly one quarter of patients, who received midostaurin, was refractory to induction therapy and relapse rate at 2 years excited 40%. Thus, new treatment options are urgently needed, particularly in r/r-AML with FLT3-ITD.

The oral second-generation bis-aryl urea tyrosine kinase inhibitor quizartinib is very specific for FLT3, has a high capacity for sustained FLT3 inhibition and an acceptable toxicity profile. Furthermore, single agent quizartinib doubled the response rate as compared to standard of care in a randomized study in r/r-AML. Although survival was also improved in this study the difference was only marginal.

In this protocol we evaluate the efficacy of quizartinib in combination with HAM (high-dose cytarabine, mitoxantrone) as compared to historical controls based on the matched threshold crossing approach followed by randomized prophylactic versus MRD-triggered continuation therapy with quizartinib including consolidation (chemotherapy as well as allo-HCT) and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myeloid leukemia according to the 2016 WHO classification (except acute promyelocytic leukemia) who are either A) refractory to induction therapy or B) relapsed after first line treatment including chemotherapy, autologous and/or allo-HCT (details below).
* Positive for FLT3-ITD (defined as a ratio of mutant to wild-type alleles of at least 0.05; measured within 2 weeks before inclusion)
* ECOG performance status ≤ 2. See appendix 18.1
* Adequate renal function defined as creatinine clearance >50 mL/min (calculated using the standard method for the institution)
* Discontinuation of prior AML treatment for at least A) 10 days for cytotoxic agents and B) 28 days for investigational drug treatment before the start of study treatment (except hydroxyurea or other treatment to control hyperleukocytosis)
* Age ≥ 18 years, no upper age limit
* Pregnancy and childbearing potential:

A) Non-pregnant and non-nursing women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).

B) Female patients of reproductive age must agree to avoid getting pregnant while on therapy.

C) WOCBP must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy) during study and 6 months after end of study/treatment. Hormonal contraception is an inadequate method of birth control.

D) Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child during study and 6 months after end of study/treatment

* Signed written informed consent
* Ability of patient to understand character and consequences of the clinical trial
* Refractory to induction therapy is defined as no CR, or CRi, or PR (according to standard criteria) [1] after 1 or 2 intensive induction cycles of at least 7 days of cytarabine 100-200mg/m² continuously or an equivalent regimen with cytarabine with total dose not less than 700mg/m² per cycle and 2 days of an anthracycline (e.g. daunorubicin, idarubicin).
* Relapsed after first line therapy is defined as relapsed AML (according to standard criteria) [1] after a first line therapy including at least one intensive induction and consolidation therapy including (but not limited to) allo-HCT.

Exclusion Criteria:

* Acute promyelocytic leukemia (AML FAB M3 with t(15;17)(q22;q12) / PML-RARA)
* Patients with known CNS leukemia
* Isolated extramedullary manifestation of AML
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy for more than one year and are considered by their physician to be at less than 30% risk of relapse within one year
* Hyperleukocytosis (leukocytes > 30,000/µl) at the time of study entry. 1)
* Uncontrolled or significant cardiovascular disease, including any of the following:

  * History of heart failure NYHA class 3 or 4
  * Left ventricular ejection fraction (LVEF) ≤ 40% by echocardiogram (ECHO)
  * History of uncontrolled angina pectoris or myocardial infarction within 12 months prior to screening
  * History of second (Mobitz II) or third degree heart block or any cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Inadequate liver function: ALT and AST ≥ 2.5 x ULN), total bilirubin ≥ 1.5 x ULN; Alkaline phosphatase ≥ 2.5 x ULN. Known liver cirrhosis or history of veno-occlusive disease (VOD) or history of Sinusoidal Obstruction Syndrome (SOS)
* Known positivity for HIV, active HBV, HCV or hepatitis A infection (active hepatitis B defined by HBs Ag positivity, active hepatitis C defined by positive virus load)
* Uncontrolled active infection
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
* within 100 days after allo-HCTat the time of screening
* clinically relevant Graft-versus-Host-Disease (GvHD) requiring initiation of treatment or treatment escalation within 21 days prior to screening
* Any one of the following ongoing or in the previous 6 months: myocardial infarction, congenital long QT syndrome, Torsades de pointes, arrhythmias (including sustained ventricular tachyarrhythmia), right or left bundle branch block and bifascicular block, unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism; as well as bradycardia defined as <50 bpms
* QTc interval >470 msec using the Fredericia correction (QTcF).
* Patients known to be refractory to platelet or packed red cell transfusions as per institutional guidelines, or who are known to refuse or who are likely to refuse blood product support.
* Severe neurologic or psychiatric disorder interfering with ability of giving informed consent
* Known or suspected active alcohol or drug abuse
* No consent for biobanking and for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation.
* Pregnancy and lactation
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Prior treatment with quizartinib

  1. These patients should be treated with hydroxyurea and / or receive leukocytapheresis treatment according to routine practice and are only allowed to enter into the study when leukocyte counts of 30,000/µl or below are reached. If hydroxyurea is not sufficient to control hyperleukocytosis, i.v. application of 100mg cytarabine continuously over 24 hours may be discussed with the Principle Investigator or the Medical Coordinator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
CRR | Collected during the first MRD-analysis / after approximately 100 study days
  Composite remission rate defined as the proportion of patients experiencing a CR (Complete remission)/CRi (Complete remission with incomplete hematological recovery rate) after salvage therapy.

SECONDARY OUTCOMES:
EFS | Collected at a minimum at baseline, day 22 of Salvage therapy, last day of second cycle of consolidation therapy, 3-monthly during maintenance therapy, at EOT, 3-monthly during FU, and yearly after 2 years during FU, at EOS
  Event-free survival
RFS | Collected at a minimum at baseline, day 22 of Salvage therapy, last day of second cycle of consolidation therapy, 3-monthly during maintenance therapy, at EOT, 3-monthly during FU, and yearly after 2 years during FU, at EOS
  Relapse-free survival
OS | Collected at a minimum at baseline, day 22 of Salvage therapy, last day of second cycle of consolidation therapy, 3-monthly during maintenance therapy, at EOT, 3-monthly during FU, and yearly after 2 years during FU, at EOS
  Overall survival
CIR | Collected at a minimum at baseline, day 22 of Salvage therapy, last day of second cycle of consolidation therapy, 3-monthly during maintenance therapy, at EOT, 3-monthly during FU, and yearly after 2 years during FU, at EOS
  Cumulative incidence of relapse
CID | Collected at a minimum at baseline, day 22 of Salvage therapy, last day of second cycle of consolidation therapy, 3-monthly during maintenance therapy, at EOT, 3-monthly during FU, and yearly after 2 years during FU, at EOS
  Cumulative incidence of deaths
QoL | Collected at baseline, day 22 of Salvage therapy, last day of second cycle of consolidation therapy, 3-monthly during maintenance therapy, at EOT, 3-monthly during FU, and yearly after 2 years during FU, at EOS
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Schlenk, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg Med5, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Jaramillo S, Le Cornet L, Kratzmann M, Krisam J, Gorner M, Hanel M, Rollig C, Wass M, Scholl S, Ringhoffer M, Reichart A, Steffen B, Kayser S, Mikesch JH, Schaefer-Eckart K, Schubert J, Geer T, Martin S, Kieser M, Sauer T, Kriegsmann K, Hundemer M, Serve H, Bornhauser M, Muller-Tidow C, Schlenk RF. Q-HAM: a multicenter upfront randomized phase II trial of quizartinib and high-dose Ara-C plus mitoxantrone in relapsed/refractory AML with FLT3-ITD. Trials. 2023 Sep 15;24(1):591. doi: 10.1186/s13063-023-07421-x. PMID 37715270